CLINICAL TRIAL: NCT04226053
Title: Comprehensive Early Childhood Parenting Supports and Children's Health and Development
Brief Title: Room to Grow Evaluation for Children
Acronym: RTG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Chris Wimer, Senior Research Scientist, Columbia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AAAR1340; P2CHD058486 (NIH)
Record Dates: First submitted 2020-01-09; First posted 2020-01-13 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Parenting; Child Development
Keywords: Poverty; Children; Social support; Practical support
MeSH Terms: interventions — Child Development

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Experimental): The treatment group will consist of 160 mothers who were randomly selected to receive Room to Grow services, which include three years of social and practical support for the mother and baby through a combination of one-on-one sessions with an expert clinical social worker in-person every three months and provision of essential baby items and equipment.
  Interventions: Other: Parenting, Child Development
- Control Group (No Intervention): The control group will consist of 160 mothers who will not receive Room to Grow services.

INTERVENTIONS:
Other: Parenting, Child Development — The treatment group will consist of mothers that were randomly selected to receive Room to Grow services, which include three years of social and practical support for the mother and baby. The research-informed program model combines tailored, one-on-one sessions with an expert clinical social worker in-person every three months, provision of essential baby items including books, toys, clothing, and equipment (retail value of in-kind items over three years averages $10,000), and connections to vital community resources (e.g., housing, entitlements, child care, social services).
  Arms: Intervention Group

SUMMARY:
This research project is a small-scale randomized controlled trial (RCT) of an innovative program based in New York City called Room to Grow (RtG). Room to Grow's mission is to enrich the lives of babies born into poverty throughout their critical first three years of development. The research-informed program model combines tailored, one-on-one sessions with an expert clinical social worker in-person every three months plus ongoing communication (via phone and email), provision of essential baby items, and connections to vital community resources. The goal of Room to Grow's innovative program is to help parents increase the probability that their children will enter school ready to learn and continue on to meet their full potential in education, work, and citizenship. The therapeutic, psychodynamic approach and robust three-year long relationship with families is designed to act as the catalyst for sustainable, long-term change in parenting methods and family system stability. Critically, and in contrast to other programs aimed at improving parenting and child development, Room to Grow believes that providing concrete material assistance enhances the effectiveness of counseling and referrals to low-income families by reducing economic stress and freeing up scarce resources.

DETAILED DESCRIPTION:
The goal of RtG's innovative program is to help parents increase the probability that their children will enter school ready to learn and continue on to meet their full potential in education, work, and citizenship. The therapeutic, psychodynamic approach and robust three-year long relationship with families is designed to act as the catalyst for sustainable, long-term change in parenting methods and family system stability. Critically, and in contrast to other programs aimed at improving parenting and child development, RtG believes that providing concrete material assistance enhances the effectiveness of counseling and referrals to low-income families by reducing economic stress and freeing up scarce resources. The program builds on decades of research on the importance of parenting supports for low-income families and their children, the significance of concrete material support and poverty reduction in enhancing children's health and development, and the recognition that the early years are an effective time to provide critical supports that influence long-term outcomes. Numerous programs, such as home-visiting models that provide parenting supports to low-income new mothers have shown promising results. After decades of correlational research establishing relationships between income, poverty, and children's health and development, there is an emerging literature providing convincing causal evidence that income matters for child outcomes. Both strains of this research build upon additional research that clearly suggests early childhood is a key period of vulnerability where interventions can make a lasting difference in the fortunes of low-income children and their families. The research will build upon this literature, by testing an intervention that combines both parenting supports and meaningful provision of material support - in essence, assessing whether a combined approach can prove potentially more powerful than the sum of its parts.

The evaluation of RtG provides the unprecedented opportunity to test the combined value of parenting education with social and material supports. The project leverages an innovative approach that combines income supports, parenting education and connection to community services to promote the early health and development of young children. Both parenting and income support programs each aim to promote low- and moderate income families' positive health and development, but too often they work in isolation, potentially limiting their ability to reduce disparities in both parents' and children's health and development. RtG's innovative model provides an opportunity to test the combined effect of these services, and provide valuable information to practitioners and policy makers on the synergistic effects of these program components. The proposed research can facilitate change in the early childhood field by demonstrating preliminary evidence that this innovative model can achieve demonstrable effects on key proximal outcomes over the first year of life and provide a first step towards building the evidence for multi-pronged approaches to meeting the needs of low-income families. Findings from this study may guide the field towards more integrated approaches that combines material support, connection to resources, and parenting assistance to make real impacts in the health and development of young children. Room to Grow and its evaluation will provide clear contributions to the development of a culture of health and relevant policies in the early childhood space. This will be the first RCT that provides a combination of parenting and community supports with substantial and empowering provision of material support. Many parenting programs provide some developmentally appropriate books or toys, but it is incredibly rare to provide the retail equivalent of roughly $10,000 in support over the first three years of life. This will establish whether a model such as RtG's holds promise for transforming early childhood parenting programs in helping to build a culture of health and for reducing health disparities among children from divergent backgrounds. The organization and its leadership look forward to learning from the evaluation project in order to understand more about what's working well and what could be improved in the program delivery and curriculum. The team at RtG has purposefully created a culture that uses data to inform decision-making and looks forward to understanding the full scope of results from the RCT. RtG is currently developing plans for expansion over the next five years as part of a formal strategic planning process. The organization hopes to eventually serve double or more the number of families in each city where it operates, New York and Boston. Findings to date from internal evaluations are extremely encouraging. It is the researchers' hope that other foundations and government agencies (or private donors) will be excited to build upon support from the Robert Wood Johnson Foundation and that the researchers will be able to extend the initial momentum generated by this project over time.

The project is designed to investigate proximal outcomes. Over the long-term, the research team hopes to build upon these proximal outcomes and to eventually follow children through school-age, as well as greatly expand the number of children that are included in the RCT project.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Must be at least 16 years old
* In third trimester (weeks 28-34) of pregnancy
* Meet Room to Grow program criteria
* Low-Income
* In need of services

Exclusion Criteria:

* Cannot read/write English and/or Spanish
* Male
* Past third trimester
* Already given birth
* Mid to high income

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 322 (Actual)
Dates: Start 2017-01-13 (Actual); Primary Completion 2023-10-04 (Actual); Study Completion 2023-10-04 (Actual)

PRIMARY OUTCOMES:
Change in Mean Score of Depressive Symptoms using the CES-D Scale | At Baseline (weeks 28-34 of pregnancy); 10.5 months after birth of child; 25 months after birth of child
  The Center for Epidemiological Studies-Depression (CES-D), is a 20-item measure that asks caregivers to rate how often over the past week they experienced symptoms associated with depression, such as restless sleep, poor appetite, and feeling lonely. Response options range from 0 to 3 for each item (0 = Rarely or None of the Time, 1 = Some or Little of the Time, 2 = Moderately or Much of the time, 3 = Most or Almost All the Time). Scores range from 0 to 60, with high scores indicating greater depressive symptoms.
Change in Mean Score of Perceived Stress Scale (PSS) | At Baseline (weeks 28-34 of pregnancy); 10.5 months after birth of child; 25 months after birth of child
  The Perceived Stress Scale (PSS) is a widely used instrument for measuring the perception of general stress. This 14-item scale measures how stressful or uncontrollable participants find their lives. Respondents rate the frequency of their feelings and thoughts related to events and situations that occurred in the last month. Individual scores on the PSS can range from 0-40 with higher scores indicating higher perceived stress. Scores ranging from 0-13 would be considered low stress. Scores ranging from 14-26 would be considered moderate stress. Scores ranging from 27-40 would be considered high perceived stress.
Change in Mean Score of Parental Sense of Competence using PSOC Scale | At Baseline (weeks 28-34 of pregnancy); 10.5 months after birth of child; 25 months after birth of child
  The Parenting Sense of Competence Scale (PSOC). The PSOC measures parental competence on two dimensions: Satisfaction and Efficacy. It is a 17-item Likert-scale questionnaire (on a 6 point scale ranging from strongly agree [1] to strongly disagree [6]), with nine questions under Satisfaction and seven under Efficacy. Satisfaction section examines the parents' anxiety, motivation and frustration, while the Efficacy section looks at the parents' competence, capability levels, and problem-solving abilities in their parental role. A higher score indicates a higher parenting sense of competency.
Change in Mean Score of the Confusion, Hubbub, and Order Scale (CHAOS) | At Baseline (weeks 28-34 of pregnancy); 10.5 months after birth of child; 25 months after birth of child
  The Confusion, Hubbub, and Order Scale (CHAOS) is a questionnaire filled out by parents that is designed to assess the level of confusion and disorganization in the child's home environment. The statements are scored using a 4-point scoring system. The questionnaire consists of 15 statements, to each of which a parent or caregiver assigns a number between 1 and 4 that correspond to the following: 1 = Very much like your own home; 2 = Somewhat like your own home; 3 = A little bit like your own home; 4 = Not at all like your own home. Two items (6 and 10) from the CHAOS scale are included in the survey. A higher score represents characteristics of a more chaotic, disorganized, and hurried home. The higher the score, the more chaotic a home is considered to be.
Change in Mean Score of Cognitive Stimulation in the Home (STIMQ) | At Baseline (weeks 28-34 of pregnancy); 10.5 months after birth of child; 25 months after birth of child
  A measure of cognitive stimulation in the home consisting of 4 subscales: Availability of Learning Materials (ALM), Reading, Parental Involvement in Developmental Advance (PIDA), and Parental Verbal Responsivity (PVR). Respondents answer "Yes" or "No" in subscales and subtotals are tallied. For the ALM scale score section: 0-1: enter 0, 2-4: enter 1; 5+: enter 2 (minimum score: 0, maximum score: 8). Calculation of reading scale score includes number of books; 0: enter 0; 1-9: enter 1; 10-24: enter 2; 25-49: enter 3; 50+: enter 4 and number of days reads book each week; 0-1: enter 0; 2-3: enter 1; 4+: enter 2 (minimum score: 0, maximum score: 6). PIDA scale: questions 1-15 (minimum score: 0, maximum score: 15) and PVR questions 1-7 (minimum score: 0, maximum score: 7). Calculation of total StimQ score is the grand total of each subscale combined (maximum of 36 for four subscale totals combined). A higher score reflects greater stimulation in home (favorable).
Change in Mean Score of Aggravation in Parenting Scale | At Baseline (weeks 28-34 of pregnancy); 10.5 months after birth of child; 25 months after birth of child
  A measurement of stress experienced by parents associated with caring for children. It measures the amount of parenting stress brought on by changes in employment, income or other factors in the parent's life. Research has shown that high levels of aggravation in parenting are related to mothers' employment status and to child behavior problems. High stress and aggravation in parents are associated with poor cognitive and socioemotional development of young children. At the 10.5 month follow-up, we are using 6 of the 9 items in this scale. Response categories being (1) Strongly agree, (2) Somewhat agree, (3) Somewhat disagree, (4) Strongly disagree. This 1-4 score is reverse coded, and items are averaged to create an overall score with higher scores indicating more stress.
Number of Toys and Goods in the Home | At Baseline (weeks 28-34 of pregnancy); 10.5 months after birth of child; 25 months after birth of child
  Subjects are asked if they have certain types of developmentally appropriate toys and games in the categories of symbolic play (doll, toy pots, small car), art (crayons, Play-Doh, paint), adaptive/fine motor toys (puzzle, shape sorter, pop-up toy), language (toy letters or numbers, toys that make animal sounds) and life-size toys (toy car or animal for child to ride). Respondents can answer yes/no for each (1=yes, 0=no). A higher number (0-16 items) of developmentally appropriate toys and goods in the home reflects a more favorable outcome for the child.
Worry Enough Money for Baby | At Baseline (weeks 28-34 of pregnancy); 10.5 months after birth of child; 25 months after birth of child
  Subjects are asked to rate (on a scale of 1-10) how worried they are about having enough money to cover their baby's expenses with 1 being "Not at all worried" and 10 being "Very worried". A lower score indicates less concern and is therefore favorable.
Change in mean score of Parent Supportiveness using the 3-bag task | At follow-up in-person meeting (42-72 months after birth of child)
  The 3-bag task utilizes a semi-structured play protocol in which the parent-child dyad is instructed to play with the toys in each of three bags in a predetermined sequence. The semi-structured play interactions are videotaped and the parent-child behaviors scored in accordance with the 3-bag task coding scales used in the NICHD Study of Early Child Care. The parent supportiveness scale assesses maternal sensitivity, positive affect, and the extent to which the parent provides cognitive stimulation while interacting with their child. The coding scales included measures of both child and maternal behavior. Each scale score ranges from 1 to 7 points to indicate the prevalence and intensity of the observed domain. Scoring considers both the quantity of behavioral indicators observed and the quality or intensity of the behaviors. A score of 1 represents virtually no evidence of the particular behavior, and score of 7 indicates very high levels of the behavior.
Change in mean score of Parent Detachment using 3 bag-task | At follow-up in-person meeting (42-72 months after birth of child)
  The 3-bag task utilizes a semi-structured play protocol in which the parent-child dyad is instructed to play with the toys in each of three bags in a predetermined sequence. The semi-structured play interactions are videotaped and the parent-child behaviors scored in accordance with the 3-bag task coding scales used in the NICHD Study of Early Child Care. The parent detachment scale measures the parent's awareness of, attention to, and engagement with the child. Detachment can take the form of being consistently inattentive, being inconsistently attentive, and/or interacting with the child in a perfunctory or indifferent manner. Each scale score ranges from 1 to 7 points to indicate the prevalence and intensity of the observed domain. Scoring considers both the quantity of behavioral indicators observed and the quality or intensity of the behaviors. A score of 1 represents very low detachment, and score of 7 indicates very high detachment.
Change in Mean Score on Performance on Working Memory Span | At follow-up in-person meeting (42- 72 months after birth of child)
  This task measures working memory. Working memory involves holding information in short-term storage and attending to one item (i.e., a house) while overcoming interference from the other (i.e., an animal or color). The task requires children to perform the operation of naming and holding in mind two pieces of information simultaneously and to activate one while overcoming interference occurring from the other. The task becomes more difficult as the number of houses increases. In the pretest phase, it is established that children can name both the colors and the animals in the task. Children then receive three 1-house trials, three 2-house trials, and three 3-house trials. There are 18 items. The score on this activity is a proportion from 0 to 1, zero indicating no items correct and 1 indicating all items were correct.
Change in Mean Score on Inhibitory Motor Control Performance | At follow-up in-person meeting (42-72 months after birth of child)
  This task measures inhibitory motor control and is a standard go no-go task. Children are presented with a large green button on the screen that makes a "popping" sound when it is touched. Children are instructed to touch the button every time that they see an animal (the 'go' response) except when that animal is a pig (the 'no-go' response). No-go responses vary in difficulty depending on how many go responses preceded them. In the pretest phase, children are asked to identify all of the animals. During administration items, the task is presented in varying numbers of go trials prior to each no-go trial, including, in standard order, 1-go, 3-go, 3-go, 5-go, 1-go, 5-go, 7-go and 7-go. There are 40 items. The score on this activity is a proportion from 0 to 1, zero indicating no items correct and 1 indicating all items were correct.
Change in Mean Score on Attention Shifting Performance | At follow-up in-person meeting (42-72 months after birth of child)
  This task measures attention shifting and requires children to use flexible thinking. For the initial trials in the task, children are presented with two pictures (animals, flowers, etc.) that are similar along a single dimension of color, shape, or size. Initially, the child is explicitly told how two of the pictures are the same in some way. Then, the child is presented with a third picture alongside the original two and asked to state how the new picture is similar to one of the original pictures. This task requires the child to shift his/her attention from the initial dimension of similarity to a new dimension of similarity. In the most difficult, items all of the pictures are presented at once and children are prompted to identify both dimensions of similarity. There are 30 items. The score on this activity is a proportion from 0 to 1, zero indicating no items correct and 1 indicating all items were correct.
Change in Language Total Standard Score | At follow-up in-person meeting (42-72 months after birth of child)
  The Receptive One-Word Picture Vocabulary Test, Fourth Edition (ROWPVT-4) is a norm-referenced assessment that tests an individual's ability to match a spoken word with an image of an object, action, or concept. The test targets the ability to understand the meaning of words spoken and name what is depicted on a test plate without context. Score range 40 - 160. This is a standardized language assessment based on a mean of 100 and a standard deviation of 15. Scores of 85-115 are considered to be within the average range of functioning. Scores above 115 are considered above average and scores below 85 are considered below average. Scores from this measure indicate that a child's receptive vocabulary is above average, below average, or equivalent to their peers of the same age.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Wimer, PhD, Principal Investigator — Senior Research Scientist at CPRC, School of Social Work
Locations (1):
- Columbia University - Columbia Population Research Center (CPRC), New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Peacock S, Konrad S, Watson E, Nickel D, Muhajarine N. Effectiveness of home visiting programs on child outcomes: a systematic review. BMC Public Health. 2013 Jan 9;13:17. doi: 10.1186/1471-2458-13-17. PMID 23302300
- [Background] Duncan GJ, Morris PA, Rodrigues C. Does money really matter? Estimating impacts of family income on young children's achievement with data from random-assignment experiments. Dev Psychol. 2011 Sep;47(5):1263-79. doi: 10.1037/a0023875. PMID 21688900
- [Background] Chaudry A, Wimer C. Poverty is Not Just an Indicator: The Relationship Between Income, Poverty, and Child Well-Being. Acad Pediatr. 2016 Apr;16(3 Suppl):S23-9. doi: 10.1016/j.acap.2015.12.010. PMID 27044698
- [Background] Duncan, G.J., Magnuson, K., Kalil, A. et al. Soc Indic Res (2012) 108: 87. https://doi.org/10.1007/s11205-011-9867-9
- [Background] Cates CB, Weisleder A, Mendelsohn AL. Mitigating the Effects of Family Poverty on Early Child Development through Parenting Interventions in Primary Care. Acad Pediatr. 2016 Apr;16(3 Suppl):S112-20. doi: 10.1016/j.acap.2015.12.015. PMID 27044688
- [Background] Wimer C, Marti M, Brooks-Gunn J, Waldfogel J. Early Impacts of Room to Grow: A Multifaceted Intervention Supporting Parents and Children Age Zero to Three. Child Youth Serv Rev. 2021 Jul;126:106041. doi: 10.1016/j.childyouth.2021.106041. Epub 2021 Apr 30. PMID 34149135